CLINICAL TRIAL: NCT07108257
Title: Phase I Trial of Magnetic Resonance-Guided Focused Ultrasound (MRgFUS) Bilateral Capsulotomy for the Treatment of Refractory Bipolar Depression
Brief Title: Magnetic Resonance-Guided Focused Ultrasound Bilateral Capsulotomy for the Treatment of Refractory Bipolar Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6670
Record Dates: First submitted 2025-06-20; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: Treatment-Resistant Depression; Bipolar Depression
Keywords: TRBD; FUS; MRgFUS; capsulotomy; Focused Ultrasound; MR-guided Focused Ultrasound; refractory Bipolar Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-guided Focused Ultrasound Capsulotomy in Treatment-Resistant Bipolar Depression (Experimental): Participants in this arm will undergo MR-guided focused ultrasound (MRgFUS) capsulotomy targeting the anterior limb of the internal capsule. The procedure is intended to thermally ablate this brain region to assess safety and initial effectiveness in reducing symptoms of treatment-resistant bipolar depression (TRBD). All participants will receive the same intervention and will be followed for 24 months post-treatment to evaluate clinical outcomes, adverse events, and quality of life.
  Interventions: Device: ExAblate Neuro 4000

INTERVENTIONS:
Device: ExAblate Neuro 4000 — ExAblate Neuro 4000 is an MR-guided focused ultrasound (MRgFUS) device used to perform noninvasive thermal ablation of targeted brain tissue. In this study, ExAblate Neuro 4000 will be used to ablate the anterior limb of the internal capsule (capsulotomy) in patients with treatment-resistant bipolar depression (TRBD). The procedure is conducted under real-time MRI guidance and thermometry to assess safety and initial effectiveness in improving clinical symptoms and quality of life.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and initial effectiveness of MR-guided focused ultrasound (MRgFUS) bilateral capsulotomy in patients with treatment-resistant bipolar depression (TRBD).

DETAILED DESCRIPTION:
This study is a prospective, single arm and nonrandomized phase l study.

Participants will:

* Undergo MRgFUS capsulotomy targeting the anterior limb of the internal capsule.
* Be assessed before and after treatment for adverse events, symptom changes, and quality of life.
* Complete a battery of clinical rating scales including the Hamilton Depression Rating Scale (HAMD), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Young Mania Rating Scale (YMRS), Yale-Brown Obsessive Compulsive Scale (YBOCS), and the Columbia-Suicide Severity Rating Scale (C-SSRS), along with the Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ).

A total of 10 participants, all patients at Sunnybrook Hospital, are expected to enroll in the study. Each participant will be involved for approximately 26 months, including a 2-month pre-treatment period and 24 months of follow-up. The full study duration is estimated at 3 years, with primary results anticipated within 2 to 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 and ≤65 years of age, inclusive.
2. Patients who are competent and willing to give consent and able to attend study visits, as determined by both study Psychiatrist and the surgeon.
3. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of Bipolar Disorder, Type 1 or Type 2.
4. A minimum score of 20 on the Hamilton Depression Rating Scale (HAMD) when depressed (at least 2 weeks of major depression at the time the HAMD is conducted).
5. Treatment refractory bipolar depression indicated by at least two recommended monotherapy treatments or at least one monotherapy treatment and another combination treatment. The minimum duration for being on either of these regimens should be 4 weeks.
6. Ability to provide informed consent/competent to make medical decisions.

Exclusion Criteria:

Patients with unstable cardiac status [e.g. Unstable angina pectoris on medication, Patients with documented myocardial infarction within six months, Congestive heart failure requiring medication (other than diuretic), Patients on anti-arrhythmic drugs, Severe hypertension (diastolic BP > 100 on medication)] 2. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.

3. Laboratory biochemical evidence of abnormal bleeding and/or coagulopathy, including risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter or abnormal International Normalized Ratio) 4. Cerebrovascular disease (e.g. Cerebrovascular Accident within 6 months) or history of intracranial hemorrhage.

5. Untreated, uncontrolled sleep apnea. 6. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure.

7. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment.

8. Are participating or have participated in another clinical trial in the last 30 days.

9. Patients unable to communicate with the investigator and staff. 10. Presence of significant cognitive impairment 11. History of psychosis on clinical evaluation. 12. Catatonic or psychotic or actively suicidal on clinical evaluation. 12. Patients with brain tumors already known or revealed on pretreatment MRI. 13. Currently pregnant (as determined by history and serum Human Chorionic Gonadotropin) or lactating.

14. Chemical abuse or dependence within the previous six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-09-16 (Estimated); Study Completion 2028-07-16 (Estimated)

PRIMARY OUTCOMES:
Safety of Magnetic Resonance-guided Focused Ultrasound for patients with Treatment-Resistant Bipolar Disorder | From the treatment day visit through the 24-month post-treatment time points.
  Assessment of the frequency and severity of adverse events associated with ExAblate Transcranial Magnetic Resonance-guided Focused Ultrasound (MRgFUS) in patients with Treatment-Resistant Bipolar Disorder (TRBD). Adverse events, including procedure-related complications and neurological events, will be documented and assessed.

SECONDARY OUTCOMES:
Clinical Efficacy - Change in Depressive Symptoms Measured by the Hamilton Depression Rating Scale (HAMD-17) | Assessed at baseline, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months post-treatment.
  Evaluate the effectiveness of MR-guided Focused Ultrasound (MRgFUS) in reducing symptoms of bipolar depression. Clinical efficacy will be assessed by the change in scores on the Hamilton Depression Rating Scale - 17 item version (HAMD-17) from baseline through follow-up visits. The HAMD-17 is a clinician-administered scale that assesses the severity of depressive symptoms. Total scores range from 0 to 52, with higher scores indicating more severe depression.
Change in Depressive Symptom Severity Measured by the Beck Depression Inventory (BDI) | Assessed at baseline, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months post-treatment.
  Evaluate the effectiveness of MR-guided Focused Ultrasound (MRgFUS) in reducing depressive symptom severity using the Beck Depression Inventory, a validated patient-reported scale. Assessments will occur at baseline and at specified follow-up visits. The BDI consists of 21 items assessing symptoms of depression experienced over the past two weeks. Total scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
Clinical Efficacy - Change in Anxiety Symptoms measured by Beck Anxiety Inventory (BAI) | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment.
  Evaluate the effectiveness of MR-guided Focused Ultrasound (MRgFUS) in reducing anxiety symptom severity using the Beck Anxiety Inventory (BAI), a validated patient-reported scale. Assessments will occur at baseline and at specified follow-up visits. The BAI consists of 21 items measuring common symptoms of anxiety experienced over the past week. Each item is rated on a scale from 0 (not at all) to 3 (severely). Total scores range from 0 to 63, with higher scores indicating more severe anxiety symptoms.
Clinical Efficacy - Change in Manic Symptoms measured by Young Mania Rating Scale (YMRS) | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment.
  Evaluate the effectiveness of MR-guided Focused Ultrasound (MRgFUS) in reducing manic symptom severity using the Young Mania Rating Scale (YMRS), a validated clinician-administered rating scale. Assessments will occur at baseline and at specified follow-up visits. The YMRS consists of 11 items used to assess the severity of manic symptoms. Total scores range from 0 to 60, with higher scores indicating more severe mania.
Clinical Efficacy - Change in Obsessive-Compulsive Symptoms measured by Yale-Brown Obsessive Compulsive Scale (YBOCS) | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment
  Evaluate the effectiveness of MR-guided Focused Ultrasound (MRgFUS) in reducing obsessive-compulsive symptom severity using the Yale-Brown Obsessive Compulsive Scale (Y-BOCS). Assessments will occur at baseline and at specified follow-up visits. The Y-BOCS is a clinician-administered instrument that assesses the severity of obsessive and compulsive symptoms. Total scores range from 0 to 40, with higher scores indicating more severe obsessive-compulsive symptoms.
Change in Suicidal Ideation and Behavior measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post-treatment.
  Evaluate the effectiveness of MR-guided Focused Ultrasound (MRgFUS) in reducing suicidal ideation and behavior using the Columbia-Suicide Severity Rating Scale (C-SSRS). Assessments will occur at baseline and at specified follow-up visits. The C-SSRS is a clinician-administered tool that categorizes the severity and intensity of suicidal ideation and records the presence or absence of suicidal behavior. Suicidal ideation is rated on a scale from 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is assessed based on the occurrence of actual, aborted, or interrupted suicide attempts, and preparatory behaviors. Higher scores or presence of behaviors indicate greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No